CLINICAL TRIAL: NCT01618864
Title: Safety and Efficacy Evaluation of the Luxe™ Device for the Treatment of Facial Wrinkles and Rosacea
Brief Title: Safety and Efficacy of the Luxe Device to Treat Facial Wrinkles and Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Luxe01
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Rosacea; Wrinkles
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Luxe (Other)
  Interventions: Device: Luxe

INTERVENTIONS:
Device: Luxe — Self treatment at home in the peri-orbital and cheeks areas. Frequency: Daily treatment for 4 weeks followed by bi-weekly treatments for additional 4 weeks.

SUMMARY:
This study is designed to evaluate the efficacy and safety of the Luxe™ device for use in wrinkle and rosacea treatment.

Up to 60 subjects will treat their periorbital and cheek areas daily for 4 weeks and then twice a week for an additional 4 weeks. Evaluations of improvement will be conducted at the clinic after enrollment and during the treatment at 1, 2, 4, and 8 weeks after initiation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female between the ages of 21 and 60.
2. Non-smoker.
3. Have no prior experience with the Luxe™ device.
4. Having wrinkles, rhytides and fine lines in periorbital regions that are classified as wrinkle type 1-3 on the Crow's Feet Grading Scale and/or having rosacea cheeks regions.
5. Able and willing to comply with all visit, treatment and evaluation schedules and requirements.
6. Agree to make no changes in their existing skin-care regime, other than use of the study products, during the study period.
7. Able to understand and provide written Informed Consent.
8. Women of child-bearing age should pass a negative pregnancy test, and required to be using a reliable method of birth control at least 3 months prior to and throughout study enrollment.

Exclusion Criteria:

1. Fail to meet any of the inclusion criteria above.
2. Subject unable or unwilling to provide proper informed consent for participation.
3. Subject not able to understand the requirements of the study.
4. Pregnant or nursing women or intending to become pregnant during the course of study.
5. Reported having one of the following medical conditions that could result in potential harm to themselves or other:

   * Obvious cognitive deficit.
   * Neuromotor control difficulty with either hand.
   * Sensitivity to light.
   * History of light activated medical problems such as light triggered seizure disorders or migraine headaches.
   * Taking drugs which may cause light sensitivity.
6. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
7. Having a permanent implant in the treated area, such as metal plates and screws
8. Unable or unlikely to refrain from tanning, including the use of tanning booths, during the course of the study.
9. Prior or current skin therapy that may interfere with the evaluation of the study device: Renova, AHAs, Vitamin C, Kinerase, Tretinoin, Topical Retinoids, Topical Steroids, Antibiotics (topical or oral) within 14 days of baseline visit.

   Oral Retinoids within 6 month of baseline visit.
10. Use of oral Isotretinoin (Accutane®) within 6 months of initial treatment or during the course of the study.
11. Subject currently being treated for a dermatologic condition which may interfere with the safe evaluation of the study device (Eczema, Psoriasis, Severe sun damage, Dermatitis).
12. Patient on systemic corticosteroid therapy 6 months prior to and throughout the course of the study.
13. Subject with a history of hypersensitivity or allergy to (LED) light.
14. Subject with a history of hypersensitivity or allergy to any formulation or device component.
15. Having received a facial dermabrasion or chemical peel treatment within 3 months of treatment or during the study.
16. Prior skin treatment with laser in treated area within 3 months of initial treatment or during the course of the study.
17. Prior use of Botox, collagen, fat injections and /or other methods of skin augmentation (enhancement with injected or implanted material) in treated area within 2 month of initial treatment or during the course of the study. Treatment may not be performed, at all, over permanent dermal implants.
18. Prior ablative resurfacing procedure, brow lift, blepharoplasty or face lift in treated area with laser or other devices within 12 months of initial treatment or during the course of the study.
19. Any other surgery in treated area within 12 months of initial treatment or during the course of the study.
20. History of keloid formation or poor wound healing in a previously injured skin area.
21. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity).
22. Open laceration or abrasion of any sort on the area to be treated.
23. Active Herpes Simplex I at the time of treatment.
24. Multiple dysplastic nevi in the area to be treated.
25. Having a bleeding disorder or taking anticoagulation medications, including heavy use of aspirin, in a manner which does not allow for a minimum 10 day washout period prior to the treatment (as per the subject's physician discretion).
26. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications.
27. Having any form of active cancer (especially skin cancer: BCC, SCC, and Melanoma) at the time of enrollment and during the course of the study.
28. Significant concurrent illness, such as uncontrolled diabetes i.e. any disease state that in the opinion of the investigator would interfere with the treatment, or healing process.
29. Subjects who have initiated treatment with hormones including estrogen, progesterone, or oral contraceptives for 12 weeks or less, immediately preceding study entry, who intend to discontinue hormonal therapy during the study.
30. Participation in a study of another device or drug within 1 month prior to study enrollment or during this study, and as per the Investigator's careful discretion, as long as not contradictory to any of the above criteria.
31. Subjects with history of past or present drug/ alcohol abuse.
32. Mentally incompetent, prisoner or evidence of active substance.
33. Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sadick, MD, Principal Investigator — Sadick Dermatology; Arielle NB Kauvar, MD, Principal Investigator — New York Laser & Skin Care
Locations (2):
- United States (2):
  - New York Laser & Skin Care, New York, New York
  - Sadick Dermatology, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Luxe Treatment Group: Luxe: Self treatment at home in the peri-orbital and cheeks areas. Frequency: Daily treatment for 4 weeks followed by bi-weekly treatments for additional 4 weeks.
Period: Overall Study
Arm/Group | Luxe Treatment Group
Started | 23
Completed 2 Weeks | 19
Completed | 19 (Completed 4 weeks and 8 weeks of treatment)
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Luxe Treatment Group
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Investigator Assessment of Overall Global Aesthetic Improvement Scale (GAI)
Description: Data reported as percentage of participants showing improvement in overall score as assessed by investigator. 5 point scale of 0 (no difference) to 4 (Significantly marked improvement)provided for overall improvement in skin texture, roughness, skin color (even/blotchy), erythema and photo-damage.
Time Frame: 4, 8 weeks
Measure: Number; unit: percentage of participants
Groups:
- Luxe Treatment Group at 4 Weeks: Luxe: Self treatment at home in the peri-orbital and cheeks areas. Frequency: Daily treatment for 4 weeks followed by bi-weekly treatments for additional 4 weeks.
- Luxe Treatment Group at 8 Weeks: GAI assessment by investigator at 8 weeks.
Arm/Group | Luxe Treatment Group at 4 Weeks | Luxe Treatment Group at 8 Weeks
Number analyzed (Participants) | 19 | 19
percentage of participants | 61 | 68

2. Secondary Outcome: Subject Improvement Using the Global Aesthetic Improvement (GAI) Scale
Description: Data reported as percentage of participants showing improvement in overall score as assessed by subject. 5 point scale of 0 (no difference) to 4 (Significantly marked improvement) provided for overall improvement in skin texture, roughness, skin color (even/blotchy), erythema and photo-damage. Analogous to Outcome Measure 1.
Time Frame: 4, 8 weeks
Measure: Number; unit: percentage of participants
Groups:
- Luxe Treatment Group at 4 Weeks: Luxe: Self treatment at home in the peri-orbital and cheeks areas. Frequency: Daily treatment for 4 weeks followed by assessment.
- Luxe Treatment Group at 8 Weeks: Luxe: Self treatment at home in the peri-orbital and cheeks areas. Frequency: Daily treatment for 4 weeks followed by bi-weekly treatments for additional 4 weeks and assessment at week 8.
Arm/Group | Luxe Treatment Group at 4 Weeks | Luxe Treatment Group at 8 Weeks
Number analyzed (Participants) | 19 | 19
percentage of participants | 68 | 68

3. Secondary Outcome: Reduction in Rosacea by the Study Investigator Using a Validated Scale
Description: Data reported as percentage of participants showing improvement in rosacea scale: 4 point scale for presence of rosacea features from 0 (absent) to 3 (severe) for: flushing, nontransient erythema, papules and pustules and telangiectasia.
Time Frame: 4, 8 weeks
Population: Not all subjects had rosacea. 11 subjects evaluated at baseline and 4 weeks; 9 subjects evaluated at 8 weeks, since 2 subjects lost to follow-up.
Measure: Number; unit: percentage of participants
Groups:
- Luxe Treatment Group at 4 Weeks: Subjects with rosacea were evaluated by the investigator and a score provided according to a validated rosacea scale for improvement in features of rosacea such as flushing.
- Luxe Treatment Group at 8 Weeks: Evaluation of rosacea after 8 weeks of treatment.
Arm/Group | Luxe Treatment Group at 4 Weeks | Luxe Treatment Group at 8 Weeks
Number analyzed (Participants) | 11 | 9
percentage of participants | 64 | 89

ADVERSE EVENTS:
Time Frame: Adverse event data collected during 8 weeks of treatment.
Groups:
- Treatment Group: All treated subjects were evaluated for adverse events during the study.
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 2/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=23)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) — Mild irritation with bumps or pimples on the cheeks

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed for post-marketing study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to remove all Confidential Information from any publications or presentations to protect its intellectual property rights.